CLINICAL TRIAL: NCT06145516
Title: Preoperative Sleep-promotion to Achieve Improved Postoperative Pain Control and Recovery: a Randomized, Controlled Trial
Brief Title: Promoting Sleep to Alleviate Pain - Arthroplasty
Acronym: PROSAP-A
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Dnr 2023-03976-01
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip; Insomnia; Surgery; Pain, Postoperative; Postoperative Complications
Keywords: osteoarthritis; total knee arthroplasty; total hip arthroplasty; insomnia; sleep disturbance; postoperative pain
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip; Sleep Initiation and Maintenance Disorders; Pain, Postoperative; Postoperative Complications; Osteoarthritis; Parasomnias | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive behavioral therapy for insomnia (CBT-I) (Experimental): The CBT-I treatment will be administered in self-guided digital format over 4 weeks with addition of telehealth video-consultations with a psychologist one time per week. The CBT-I will focus on sleep restriction therapy and stimulus control, which have shown the highest efficacy for sleep improvement among components typically incorporated. A booster session will be provided 1-2 weeks postoperative.
  Interventions: Behavioral: Cognitive behavioral therapy for insomnia (CBT-I)
- Sleep education therapy (SET) (Active Comparator): The sleep education therapy will be administered in self-guided digital format over 4 weeks with addition of telehealth video-consultations with a research nurse one time per week. The SET will focus on sleep physiology, different sleep disturbances and sleep hygiene measures. A booster session will be provided 1-2 weeks postoperative.
  Interventions: Behavioral: Sleep education therapy (SET)

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy for insomnia (CBT-I) — Hybrid CBT-I (self-guided digital format focusing on sleep restriction therapy and stimulus control + telehealth video-consultations with psychologist)
  Arms: Cognitive behavioral therapy for insomnia (CBT-I)
Behavioral: Sleep education therapy (SET) — Self-guided digital sleep education (sleep hygiene, sleep physiology, sleep disturbances etc) + telehealth video-consultations with research nurse
  Arms: Sleep education therapy (SET)

SUMMARY:
PROSAP-A is a perioperative randomized, controlled trial with a 12-month follow-up period after total knee arthroplasty (TKA) or total hip arthroplasty (THA), aiming to investigate both acute and long-term postoperative effects of preoperative sleep-promotion. Participants with clinically significant insomnia symptoms will be randomized to a brief, hybrid version of cognitive behavioral therapy for insomnia (CBT-I) or sleep education therapy, administered over a 4-week period, prior to surgery. The primary objective is to evaluate effects of preoperative sleep-promotion on acute postoperative pain control. Secondary objectives include evaluation of postoperative sleep, recovery, mental health, cognitive function and alterations in blood biomarkers.

DETAILED DESCRIPTION:
Although preoperative sleep disturbance is associated with poorer acute postoperative pain control, as well as development of chronic postsurgical pain, only very limited attempts have been made to target preoperative sleep to achieve improved postoperative outcomes. This study addresses two chronic pain populations, TKA and THA patients, that suffer severely due to both sleep disturbance and painful symptoms. Patients who meet eligibility criteria, including insomnia severity index score >10 and confirmed DSM-V criteria for persistent insomnia disorder, will be randomized to a brief, hybrid version of CBT-I or sleep education therapy over a 4-week period, before surgery. The CBT-I will focus on the two components which have shown the highest efficacy for sleep improvement, sleep restriction therapy and stimulus control. The CBT-I treatment will be administered in self-guided digital format with addition of telehealth video-consultations with a psychologist one time per week. The sleep education therapy will also be provided in a hybrid format, including digital sessions and video-consultations with a research nurse. There will also be a booster session 1-2 weeks postoperative for both interventions. Participants will be carefully evaluated during on-site visits two times preoperative, pre- and post-intervention, and one time 6 months postoperative. During on-site visits, participants will complete multiple questionnaires (covering pain, pain catastrophizing, mental health, physical function, activity etc), undergo digital cognitive testing, quantitative sensory testing (QST, to determine pain detection thresholds to different stimuli, assess temporal summation, pain inhibitory capacity), provide blood samples, and initiate actigraphy (objective assessment of sleep continuity measures). In addition to the on-site visits, participants will complete questionnaires remotely 3 and 12 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* insomnia severity index score >10
* fulfill DSM-V criteria for persistent insomnia disorder
* average pain numerical rating scale (NRS) score ≥4 (scale 0 - 10) and/or movement-related pain NRS score ≥4 after 5 minutes walking
* scheduled to undergo primary (first-time, i.e., not revision surgery) TKA or THA due to osteoarthritis

Exclusion Criteria:

* uncontrolled medical disorders
* nightshift work
* ongoing major depressive disorder, bipolar disorder, psychotic disorder, substance dependence
* current history or high likelihood of primary sleep disorders (other than insomnia), including obstructive sleep apnea syndrome, narcolepsy, nocturnal myoclonus
* severely impaired vision (precluding ability to take part of study interventions)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2029-12-01 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Acute postoperative pain intensity | First 7 postoperative days
  Average pain intensity (NRS 0 - 10) over the past 24 h rated each morning, averaged over 7 days

SECONDARY OUTCOMES:
Pre- and acute postoperative change in sleep measures from baseline | Up to 2 weeks postoperative
  insomnia severity index, Pittsburgh sleep quality index, actigraphic sleep continuity measures (sleep onset latency, total sleep time, wakefulness after sleep onset, sleep efficiency)
Acute postoperative opioid consumption | Postoperative day (POD) 1 and POD1-7
  Oral morphine mg equivalents (OMEQs)
Recovery in the acute postoperative phase | First 7 postoperative days
  Quality of recovery (QoR) 15 score
Long-term postoperative sleep quality | Up to 12 months postoperative
  insomnia severity index
Postoperative objective sleep continuity | Up to 6 months postoperative
  actigraphic sleep efficiency [SE]
Pain intensity 6 months postoperative | 6 months postoperative
  Average pain intensity (NRS 0 - 10) over the past 24 h rated each morning, averaged over 7 days
Change in pain measures from baseline | Up to 12 months postoperative
  BPI pain severity and pain interference score, QoR-15 pain score, WOMAC OA pain score
Changes in quantitative sensory testing (QST) measures of pain | Up to 6 months postoperative
  Pressure pain threshold, temporal summation, conditioned pain modulation, cold pressor test
Change in cognitive function | Up to 6 months postoperative
  Digital cognitive testing (Mindmore platform) incl. memory, attention and processing speed, executive functions
Change in anxiety from baseline | Up to 6 months postoperative
  Generalized anxiety disorder 7 (GAD-7) score
Change in depression from baseline | Up to 6 months postoperative
  Patient health questionnaire 9 (PHQ-9) score
Change in quality of life | Up to 6 months postoperative
  EuroQol 5 dimension 5 level (EQ-5D-5L), RAND-36
Change in health-related function | Up to 6 months postoperative
  EQ-5D-5L, RAND-36
Change in osteoarthritis-related symptoms | Up to 12 months postoperative
  WOMAC OA

OTHER OUTCOMES:
Change in physical activity | Up to 6 months postoperative
  International physical activity questionnaire short form (IPAQ-sf)
Change in pain catastrophizing | Up to 6 months postoperative
  Pain catastrophizing scale (PCS)
Change in kinesiophobia | Up to 6 months postoperative
  Tampa scale of kinesiophobia (TSK)
Change in subjective pain sensitivity | Up to 6 months postoperative
  Pain sensitivity questionnaire (PSQ)
Fibromyalgia severity score | Up to 6 months postoperative
  Sum of widespread pain index + symptom severity scale (ACR 2016)
Pain-related acceptance | Up to 6 months postoperative
  Chronic pain acceptance questionnaire (CPAQ-8)
Changes in blood biomarkers | Up to 6 months postoperative
  Inflammatory mediators, monoamine metabolites, coagulation system etc

CONTACTS AND LOCATIONS:
Overall Officials: Martin F Bjurström, MD, PhD, Principal Investigator — Uppsala University / Uppsala University Hospital
Locations (1):
- Department of Surgical Sciences, Uppsala University, Uppsala, Uppland, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bjurstrom MF, Bothelius K, Maathz P, Jernelov S, Kraepelien M, Rosenstrom AHC, Niklasson A, Smith MT, Olmstead R, Irwin MR, Finan PH, Kosek E. Randomised, controlled clinical trial evaluating the effects of preoperative insomnia treatment on postoperative pain control and recovery: a protocol for the Promoting Sleep to Alleviate Pain-Arthroplasty (PROSAP-A) trial. BMJ Open. 2025 Jul 30;15(7):e099785. doi: 10.1136/bmjopen-2025-099785. PMID 40738630